CLINICAL TRIAL: NCT04656821
Title: Ultrasound Guided Erector Spinae Block Versus Ultrasound Guided Thoracic Paravertebral Block for Pain Relief in Patients With Acute Thoracic Herpes Zoster
Brief Title: Erector Spinae Block Versus Thoracic Paravertebral Block for Acute Thoracic Herpes Zoster
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Esraa Hassan Abdelwahab, Assistant lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32720/11/18
Record Dates: First submitted 2020-12-04; First posted 2020-12-07 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Acute Thoracic Herpes Zoster; Erector Spinae Plane Block; Thoracic Paravertebral Block; Pain Relief
MeSH Terms: interventions — Tin Fluorides

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): Patients of this group will receive standard treatment for herpes zoster which include acyclovir 800 mg, 5 times daily administered orally within the first 72 hours and analgesics as needed.
  Interventions: Drug: Control Rx
- Erector Spinae Block (ESB) group (Experimental): Patients of this group will receive 25 mg bupivacaine 0.5%, plus 8 mg dexamethasone in a total volume of 10 ml (The final Patients of this group will receive 25 mg bupivacaine 0.5%, plus 8 mg dexamethasone in a total volume of 10 ml(The final concentration of bupivacaine will be 0.25%) to be injected beneath the erector spinae muscle sheath) at the desired level under ultrasonography. The concentration of bupivacaine will be 0.25%) to be injected beneath the erector spinae muscle sheath) at the desired level under ultrasonography.
  Interventions: Procedure: Erector Spinae Block
- Thoracic Paravertebral Block group (Experimental): Patients will receive 25 mg bupivacaine 0.5%, plus 8mg dexamethasone in a total volume of 10 ml(The final concentration of bupivacaine will be 0.25%) to be injected in the Paravertebral space at the desired level under ultrasonography
  Interventions: Procedure: Thoracic Paravertebral Block

INTERVENTIONS:
Drug: Control Rx — Patients of this group will receive standard treatment for herpes zoster which include acyclovir 800 mg, 5 times daily administered orally within the first 72 hours and analgesics as needed
  Arms: Control Group
Procedure: Erector Spinae Block — Patients of this group will receive 25 mg bupivacaine 0.5%, plus 8 mg dexamethasone in a total volume of 10 ml (The final concentration of bupivacaine will be 0.25%) to be injected beneath the erector spinae muscle sheath) at the desired level under ultrasonography.
  Arms: Erector Spinae Block (ESB) group
Procedure: Thoracic Paravertebral Block — Patients of this group will receive 25 mg bupivacaine 0.5% , plus 8mg dexamethasone in a total volume of 10 ml(The final concentration of bupivacaine will be 0.25%) to be injected in the Paravertebral space at desired level under ultrasonography
  Arms: Thoracic Paravertebral Block group

SUMMARY:
The aim of this research is to study and compare the efficacy and safety of single injection erector spinae plane block and thoracic paravertebral block in prevention of post herpetic neuralgia in patients with acute thoracic herpes zoster.

ELIGIBILITY:
Inclusion Criteria:

* Over 50 years of age
* Chest wall herpetic eruption of less than one week
* Moderate or severe pain

Exclusion Criteria:

* Patient refusal
* Eruption more than one week duration
* Patients who will not receive appropriate anti-viral therapy
* Patients with mild pain
* Infection at the site of injection
* Patients with a history of renal, hepatic diseases, coagulopathy, steroid therapy, malignancies.
* Patient taking chemotherapy and/or radiotherapy.

Ages: 51 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-12-05 (Actual); Primary Completion 2021-06-06 (Estimated); Study Completion 2021-06-20 (Estimated)

PRIMARY OUTCOMES:
The incidence of post herpetic neuralgia (PHN) | 3 months
  Persistent herpetic pain after 3 months will reported as post herpetic neuralgia (PHN)

SECONDARY OUTCOMES:
Visual Analog Scale | 6 months
  Visual Analog Scale (VAS) at baseline, 3, 4, 12, 24 weeks
Total consumption of rescue analgesia | 6 months
  Rescue analgesia in the form of Acetaminophen in a dose of 1,000 mg will be given if Visual Analog Scale (VAS) ≥4
The times of complete resolution of pain | 3 months
  The times of complete resolution of pain (from the date of block until complete disappearance of herpetic pain)
Adverse effects and complications | 1 day
  * Hypotension
  * Pneumothorax
  * Local anesthetic toxicity
  * Respiratory depression

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request
Supporting Information: Study Protocol, SAP